CLINICAL TRIAL: NCT00110929
Title: A Study to Compare the Efficacy and Safety of an Oral Calcimimetic Agent (AMG 073) When Two Different Vitamin D Regimens Are Used in Subjects With Secondary Hyperparathyroidism of End-Stage Renal Disease (ESRD)
Brief Title: Treatment for Patients With Secondary Hyperparathyroidism of End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020158
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: End Stage Renal Disease
Keywords: Sensipar®; Secondary HPT; Mimpara®; Cinacalcet; calcimimetic; End-Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cinacalcet

INTERVENTIONS:
Drug: AMG 073

SUMMARY:
The purpose of this research is to study the efficacy and safety of AMG 073 in patients with kidney failure who are being treated with hemodialysis or peritoneal dialysis and who also have secondary hyperparathyroidism (HPT).

ELIGIBILITY:
Inclusion Criteria: - Completed one of the qualifying studies (i.e., patient previously took part in an Amgen study investigating the drug AMG 073 and its effects on secondary hyperparathyroidism [HPT]; in particular parathyroid hormone [PTH], calcium and phosphorus levels in blood associated with kidney failure) - Must agree to use, in the opinion of the principal investigator, highly effective contraceptive measures throughout the study Exclusion Criteria: - Pregnant or nursing females - Experienced a myocardial infarction within 3 months before day 1 - Have an unstable medical condition, defined as having been hospitalized, other than for dialysis vascular access revision, within 30 days before day 1, or otherwise unstable in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850
Dates: Start 2002-11

PRIMARY OUTCOMES:
Examine PTH and Ca x P control when cinacalcet is administered in the setting of flexible dosing of vitamin D sterols.

SECONDARY OUTCOMES:
Examine safety and tolerability of cinacalcet.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Sprague SM, Evenepoel P, Curzi MP, Gonzalez MT, Husserl FE, Kopyt N, Sterling LR, Mix C, Wong G. Simultaneous control of PTH and CaxP Is sustained over three years of treatment with cinacalcet HCl. Clin J Am Soc Nephrol. 2009 Sep;4(9):1465-76. doi: 10.2215/CJN.06141108. Epub 2009 Aug 20. PMID 19696213
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20020158.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20020158.pdf